CLINICAL TRIAL: NCT03012412
Title: Mindfulness Based Program for Infertility
Acronym: MBPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Portuguese Fertility Association (Unknown)
Responsible Party: Principal Investigator, Ana Galhardo, Principal Investigator, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/68392/2010-04
Record Dates: First submitted 2016-12-30; First posted 2017-01-06 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Program for Infertility (Experimental): Behavioral: MBPI
  The Mindfulness Based Program for Infertility is a manualized group psychological intervention derived from contextual or 3rd wave cognitive-behavioral therapies intended to develop mindfulness and acceptance skills, as well as to promote perceptions of self-efficacy to deal with the demands of an infertility diagnosis and medical treatment. It comprises 10 weekly sessions of approximately 2hr each, run in small groups (ranging from 10 to 15 participants).
  Interventions: Behavioral: Mindfulness Based Program for Infertility
- Treatment As Usual (TAU) (No Intervention): Standard infertility medical treatment provided by IVF clinics (public and private) - no psychological intervention being pursued.

INTERVENTIONS:
Behavioral: Mindfulness Based Program for Infertility — The Mindfulness Based Program for Infertility is a manualized group psychological intervention derived from contextual or 3rd wave cognitive-behavioral therapies intended to develop mindfulness and acceptance skills, as well as to promote perceptions of self-efficacy to deal with the demands of an infertility diagnosis and medical treatment. It comprises 10 weekly sessions of approximately 2hr each, run in small groups (ranging from 10 to 13 participants).
  Other Names: MBPI
  Arms: Mindfulness Based Program for Infertility

SUMMARY:
The current study aims to test the efficacy a mindfulness based intervention for women facing fertility problems - the Mindfulness Based Program for Infertility (MBPI). MBPI comprises 10 weekly group sessions of approximately 2 hours each, run in small groups of 10-15 women. The main goal of MBPI intervention is to reduce depressive and anxiety symptoms and promote infertility self-efficacy and acceptance and mindfulness skills. The MBPI is intended to develop willingness/acceptance through a process of contacting the present moment and be in touch with the unfolding experience in an open and non-judgmental way, particularly infertility-related experiences.

DETAILED DESCRIPTION:
The Mindfulness Based Program for Infertility (MBPI) was developed based on the Mindfulness Based Program for Stress Reduction, the Mind/Body Program for Infertility and basic principles of Acceptance and Commitment Therapy. This program aims, fundamentally, learning and practicing emotion regulation skills, particularly mindfulness and acceptance. It addresses values (chosen life directions) clarification, interpersonal communication, healthy lifestyles, and emotional self-care. The training of these skills occurs at all sessions and is also encouraged between sessions. Support materials are provided for this, including a Participant's Manual and an audio CD with several mindfulness meditation instructions. The MBPI encloses 10 weekly sessions of 2 hours each, except for one of the sessions that lasts for one day. It is a structured psychosocial intervention program, with a group format (max. 15 women). Male partners are invited to participate in 3 sessions.

MBPI sessions were carried out by a clinical psychologist with previous training in contextual-behavioral therapies. A Therapist Manual was structured, describing the details for conducting each session.

Most of the MBPI sessions follow a similar structure. They begin with a first half-hour of sharing (optional). After the first half hour a formal mindfulness practice is held, followed by sharing how participants felt, what they have noticed, how was the experience for them. The set of formal practices selected for the MBPI is commonly used in mindfulness programs. Informal mindfulness practice is also presented as early as the second session through mindful eating. The three minutes breathing space exercise ends each session. Metaphors and experiential exercises are included in most of the sessions. These comprise an experiential exercise of listening to others, the introduction of values clarification (valued life directions) through the imagery exercise "10 years of marriage", the integration of a greater number of positive aspects in day-to-day experience, a psychoeducational component regarding healthy lifestyle (exercise, nutrition, caffeine, alcohol, nicotine, etc.). Moreover, the promotion of psychological flexibility/acceptance is intended to be achieved through mindfulness practice, but also through the use of metaphors such as "the mind as a radio always on", "the coach and passengers" and through emphasizing the importance of values clarification and committed action.

Previously to data collection, ethical approval was obtained from the Scientific Council of the Faculty of Psychology and Educational Sciences of the University of Coimbra. Participants were women aged 18 years old or older, presenting a medically established infertility diagnosis. Participants answered a recruitment announcement posted at the Portuguese Fertility Association (patients association) website after getting the approval of this association board. Participants were informed about the voluntary and confidential nature of the data. A semi-structured clinical interview was used for MBPI admission. This interview allows the gathering of demographic and clinical data and the screening for severe psychopathology. Women who answered the recruitment announcement but lived in places where the MBPI sessions were not scheduled were invited to participate in the study as members of the control group and were given the opportunity to participate in future editions.

All participants were required to sign the informed consent and a numerical unique code was assigned to each participant.

The study encompassed three different assessment moments (T0, T1, T2) namely before intervention (T0), at the end of the intervention (T1) and at six months (T2). Another follow-up study conducted seven years (T3) after the intervention was also designed for the participants who completed the MBPI (not the control group).

The assessment protocol was completed at home. It was delivered to the participants in the MBPI group during the admission interview and at the end of the last MBPI session. It was then returned to the research team by mail. The assessment protocol was sent and returned by mail to participants in the control group (stationary post envelopes were provided). Concerning the seven years follow-up study data collection was carried out online.

All quantitative data were analyzed using SPSS (version 20). Independent samples t tests were conducted to explore whether there were differences between the groups regarding demographic variables. Depending on the nature of clinical variables, the groups were compared through independent samples t tests, qui-squared tests and Fisher tests. When significant differences were found Pearson and point-biserial correlation coefficients were used. Independent samples t tests were also performed to explore the equivalence between the groups regarding the study variables. The effect size considered for these analyses was the Eta square (ƞ2).

To explore mean differences between pre-treatment (T0) and post-treatment (T1) (main time effect), between groups (main group effect) and time X group interaction effect repeated measures ANOVAs were conducted, considering the MBPI and the control group as the between-subjects factor. Mean differences of the study variables were also studied in each group through paired samples t tests. In order to explore mean differences between post-treatment (T1), six-months follow-up (T2) and 7 years follow-up (T3) in MBPI participants repeated measures ANOVAs were conducted. Effect sizes were assessed through partial Eta2 (ƞ2p). Independent samples t tests and repeated measures ANOVAs assumptions were verified through Skweness and Kurtosis measures. Sphericity assumption for the repeated measures ANOVAs were analyzed through Mauchly's W. Whenever this assumption was not verified we used the Huynh-Feldt Epsilon (ɛ > .75) or the Greenhouse-Geisser Epsilon (ɛ < .75), that correspond to probability correction factors of the F statistics significance.

Lastly, to understand mechanisms underlying the effect of the MBPI on the reduction of depressive symptoms scores, a mediation analysis based upon regression analysis was conducted. In this model, the intervention was the predictor (coded as 0 = control; 1 = MBPI), self-efficacy at T1 was the mediator variable and depressive symptoms at T1 was the outcome variable. Self-efficacy and depressive symptoms at T0 were included as covariates in the model, to allow for a better prediction model, rather than using computed variables based on the changes in these scores. Significance of indirect effects was calculated using PROCESS macro in SPSS (Model 4) with bootstrap procedures (5000 samples) for determining statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Women dealing with an infertility diagnosis (independently of female, male, both female and male or unknown factor), pursuing infertility medical treatment

Exclusion Criteria:

* Severe psychiatric problems assessed through a semi-structured clinical interview used for MBPI admission

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-05; Primary Completion 2013-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms assessed by the Beck Depressive Inventory (BDI) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Beck Depressive Inventory (BDI)
Changes in Mindfulness skills assessed by the Five Facet Mindfulness Questionnaire (FFMQ) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Five Facet Mindfulness Questionnaire (FFMQ)
Changes in perceptions of infertility self-efficacy assessed by the Infertility Self-efficacy Scale (ISE) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Infertility Self-efficacy Scale (ISE)

SECONDARY OUTCOMES:
Changes in anxiety symptoms assessed by the Spielberger State Anxiety Inventory (STAI-Y1) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Spielberger State Anxiety Inventory (STAI-Y1)
Changes in acceptance skills assessed by the Acceptance and Action Questionnaire (AAQ-II) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Acceptance and Action Questionnaire (AAQ-II)
Changes in self-compassion assessed by the Self-compassion Scale (SCS) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Self-compassion Scale (SCS)

OTHER OUTCOMES:
Changes in external shame assessed by the Others As Shamer (OAS) | 7 years and 8 months (from Baseline to 7-years follow-up)
  Assessed by the Others As Shamer (OAS)
Changes in entrapment assessed by the Entrapment Scale (ES) | 8 months (from Baseline to 6-months follow-up)
  Assessed by the Entrapment Scale (ES)
Changes in defeat assessed by the Defeat Scale (DS) | 8 months (from Baseline to 6-months follow-up)
  Assessed by the Defeat Scale (DS)

CONTACTS AND LOCATIONS:
Overall Officials: José A Pinto-Gouveia, MD, PhD, Study Chair — CINEICC - Faculty of Psychology and Educational Sciences of the University of Coimbra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galhardo A, Cunha M, Pinto-Gouveia J. Measuring self-efficacy to deal with infertility: Psychometric properties and confirmatory factor analysis of the Portuguese version of the infertility self-efficacy scale. Res Nurs Health. 2013 Feb;36(1):65-74. doi: 10.1002/nur.21516. Epub 2012 Oct 18. PMID 23081663
- [Background] Galhardo A, Moura-Ramos M, Cunha M, Pinto-Gouveia J. The infertility trap: how defeat and entrapment affect depressive symptoms. Hum Reprod. 2016 Feb;31(2):419-26. doi: 10.1093/humrep/dev311. Epub 2015 Dec 17. PMID 26677954
- [Background] Galhardo A, Pinto-Gouveia J, Cunha M, Matos M. The impact of shame and self-judgment on psychopathology in infertile patients. Hum Reprod. 2011 Sep;26(9):2408-14. doi: 10.1093/humrep/der209. Epub 2011 Jul 4. PMID 21727160
- [Result] Galhardo A, Cunha M, Pinto-Gouveia J. Mindfulness-Based Program for Infertility: efficacy study. Fertil Steril. 2013 Oct;100(4):1059-67. doi: 10.1016/j.fertnstert.2013.05.036. Epub 2013 Jun 27. PMID 23809500